CLINICAL TRIAL: NCT01654549
Title: The Effect of Helicobacter Pylori Eradication on Liver Fat Content in Non-diabetic Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Helicobacter Pylori Eradication in Non-diabetic Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Assistant professor of medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1391/3/27-573
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Steatohepatitis,; Helicobacter pylori,; Insulin resistance,; Alanine aminotransferase,; Aspartate aminotransferase,
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle modification (No Intervention): Obtaining ideal body weight by calorie restriction diet and programmed physical activity
- H.pylori eradication (Experimental): H.pylori eradication by quadruple antibiotic therapy for two weeks plus obtaining ideal body weight by calorie restriction diet and programmed physical activity
  Interventions: Drug: H.pylori eradication

INTERVENTIONS:
Drug: H.pylori eradication — Omeprazole (20 mg/BD)+ Amoxicillin (1 g/day)+ Bismuth subcitrate (240 mg/BD)+ Azithromycin (500 mg/BD)
  Other Names: H.pylori treatment
  Arms: H.pylori eradication

SUMMARY:
The aim of study was to evaluate the effect of helicobacter pylori eradication on liver fat content, liver function tests, lipid profile, homeostasis model assessment-IR (HOMA-IR) index, and anthropometric measurements (body mass index and waist circumference)in non-diabetic subjects with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) antigens have been found in the liver of individuals with benign and malignant liver diseases. The role of HP in the pathogenesis of non-alcoholic fatty liver disease (NAFLD) is controversial.

This randomized double blind clinical trial was performed in non-diabetic dyspeptic patients with positive antibody to HP and the evidence of fatty liver in ultrasonography. After excluding other causes, participants with persistent elevated serum aminotransferase levels were presumed to have NAFLD. Those with NAFLD liver fat score greater than (-0.64) and positive urea breath test (UBT) were enrolled. They were randomly assigned to lifestyle modification alone or lifestyle modification plus HP eradication groups. Quadruple therapy (omeprazole, amoxicillin, bismuth subcitrate, and clarithromycin) for HP eradication was performed in two weeks. HP eradication was documented by UBT. Liver fat content, fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein, HOMA-IR, and anthropometric measurements (body mass index and waist circumference) were checked at baseline and six weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Dyspeptic patients with positive antibody to H.pylori and persistent elevated aminotransferase levels with the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic.

Exclusion Criteria:

* Alcohol use (more than 20 gram per day in men and 10 gram per day in women per day), diabetes mellitus, heart disease (ischemic or congestive), hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion), renal disease (serum creatinine concentration of > 1.5 mg/dl), any severe systemic co-morbidities, neoplasm, using any medication during the past 3 months, previous history of peptic ulcer, previous history of H.pylori eradication, existence of alarm signs (weight loss, dysphagia, anemia, vomiting, positive family history of gastrointestinal cancers), and pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gastroenterology clinic, Sina hospital., Tehran, Iran

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Modification | H.Pylori Eradication
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — H.pylori eradication not successful | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Modification | H.Pylori Eradication | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.90 (13.96) | 41.11 (10.14) | 41.57 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Liver Fat Content
Description: Primary outcome measure was changes in the liver fat content from baseline to the end of study (6 weeks post-treatment).
  The percent of liver fat was calculated as below:
  "Liver fat content (%) = 10 (-0.805 + 0.282 * metabolic syndrome (yes = 1 / no = 0) + 0.078 * type 2 diabetes (yes =2 / no =0) + 0.525 * log fasting serum insulin (mU/L) + 0.521 * log fasting serum AST (U/L) - 0.454 * log (AST/ALT)"
Time Frame: 8 weeks (6 weeks post-treatment)
Measure: Mean (Standard Deviation); unit: percentage of liver fat content
Groups:
- Liver Fat Content in H.Pylori Eradication at Baseline: Liver fat content in Helicobacter pylori eradication plus lifestyle modification group at baseline
- Liver Fat Content in H.Pylori Eradication at 8 Weeks: Liver fat content in Helicobacter pylori eradication plus lifestyle modification group at 8 weeks
- Liver Fat Content in Lifestyle Modification at Baseline: Liver fat content in lifestyle modification group at baseline
- Liver Fat Content in Lifestyle Modification at 8 Weeks: Liver fat content in lifestyle modification group at 8 weeks
- Liver Fat Content Change in H.Pylori Eradication: The change of liver fat content from baseline to the end of study in H.pylori eradication group
- Liver Fat Content Change in Lifestyle Modification: The change of liver fat content from baseline to the end of study in lifestyle modification group
Arm/Group | Liver Fat Content in H.Pylori Eradication at Baseline | Liver Fat Content in H.Pylori Eradication at 8 Weeks | Liver Fat Content in Lifestyle Modification at Baseline | Liver Fat Content in Lifestyle Modification at 8 Weeks | Liver Fat Content Change in H.Pylori Eradication | Liver Fat Content Change in Lifestyle Modification
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 19 | 20
percentage of liver fat content | 8.38 (4.47) | 7.72 (4.34) | 8.50 (6.03) | 7.29 (5.06) | 0.66 (0.61) | 1.21 (1.31)
Statistical Analysis 1: Comparison: Liver Fat Content in H.Pylori Eradication at Baseline vs Liver Fat Content in Lifestyle Modification at Baseline; Test type: Superiority or Other; p = 0.94, t-test, 2 sided
Statistical Analysis 2: Comparison: Liver Fat Content in H.Pylori Eradication at 8 Weeks vs Liver Fat Content in Lifestyle Modification at 8 Weeks; Test type: Superiority or Other; p = 0.78, t-test, 2 sided
Statistical Analysis 3: Comparison: Liver Fat Content in H.Pylori Eradication at Baseline vs Liver Fat Content in H.Pylori Eradication at 8 Weeks; Test type: Superiority or Other; p < 0.01, Paired t-test
Statistical Analysis 4: Comparison: Liver Fat Content in Lifestyle Modification at Baseline vs Liver Fat Content in Lifestyle Modification at 8 Weeks; Test type: Superiority or Other; p < 0.01, Paired t-test
Statistical Analysis 5: Comparison: Liver Fat Content Change in H.Pylori Eradication vs Liver Fat Content Change in Lifestyle Modification; Test type: Superiority or Other; p = 0.10, t-test, 2 sided

2. Secondary Outcome: Serum Alanine Aminotransferase Level
Description: Secondary outcome measure was change in serum alanine aminotransferase concentration from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Serum Aspartate Aminotransferase Level
Description: Secondary outcome measure was change in serum aspartate aminotransferase concentration from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Fasting Serum Glucose
Description: Secondary outcome measure was change in fasting serum glucose concentration from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Serum Lipid Profile
Description: Secondary outcome measure was change in serum lipid profile (including serum triglyceride, cholesterol, low-density lipoprotein, and high-density lipoprotein concentration) from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Homeostasis Model Assessment-Insulin Resistance (HOMA-IR)
Description: Secondary outcome measure was change in HOMA-IR from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Anthropometric Measurements
Description: Secondary outcome measure was change in anthropometric measurements (body mass index and waist circumference) from baseline to the end of study
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: self-reporting by participants
Groups:
- H. Pylori Eradication: Helicobacter pylori eradication
- No Intervention: Lifestyle modification
Arm/Group | H. Pylori Eradication | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
No limitations and Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes